CLINICAL TRIAL: NCT05014828
Title: A Multicenter, Open-label, Phase 2 Study to Evaluate the Efficacy and Safety of Tislelizumab in Combination With Lenvatinib in Patients With Selected Solid Tumors
Brief Title: To Evaluate the Efficacy and Safety of Tislelizumab in Combination With Lenvatinib in Participants With Selected Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-212; CTR20211874 (Other: ChinaDrugTrials)
Record Dates: First submitted 2021-07-28; First posted 2021-08-20 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor
Keywords: Solid tumors
MeSH Terms: interventions — lenvatinib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Safety Run In (Experimental): Participants with advanced or metastatic unresectable solid tumors were enrolled to receive 400 mg of tislelizumab administered on Day 1 of each 6-week cycle, along with 20 mg of lenvatinib self-administered orally once daily, to determine the recommended Part 2 dose (RP2D).
  Interventions: Drug: lenvatinib; Drug: Tislelizumab
- Part 2: Squamous Cell Carcinoma of the Head and Neck (SCCHN) Cohort (Experimental): Participants with previously untreated, advanced or metastatic SCCHN received tislelizumab (400 mg administered intravenously [IV] every 6 weeks [Q6W]) in combination with lenvatinib (20 mg taken orally once daily [QD]) until disease progression, start of new anticancer therapy, unacceptable toxicity, withdrawal of consent, or study termination.
  Interventions: Drug: lenvatinib; Drug: Tislelizumab
- Part 2: Renal Cell Carcinoma (RCC) Cohort (Experimental): Systemic therapy naive participants with advanced or metastatic RCC received tislelizumab (400 mg IV Q6W) plus lenvatinib (20 mg orally QD) until disease progression, start of new anticancer therapy, unacceptable toxicity, withdrawal of consent, or study termination.
  Interventions: Drug: lenvatinib; Drug: Tislelizumab
- Part 2: Non-Small Cell Lung Cancer (NSCLC) Cohort (Experimental): Participants with NSCLC expressing programmed cell death-ligand 1 (PD-L1) in ≥1% of tumor cells (TC ≥1%) and who had not received prior systemic therapy received tislelizumab (400 mg IV Q6W) and lenvatinib (20 mg orally QD) until disease progression, start of new anticancer therapy, unacceptable toxicity, withdrawal of consent, or study termination; this cohort was closed early based on emerging external data.
  Interventions: Drug: lenvatinib; Drug: Tislelizumab
- Part 2: Gastric Cancer (GC) Cohort (Experimental): Participants with advanced GC who had received one prior line of systemic therapy were enrolled to receive tislelizumab and lenvatinib at the RP2D (tislelizumab 400 mg IV Q6W; lenvatinib 20 mg orally QD) until disease progression, start of new anticancer therapy, unacceptable toxicity, withdrawal of consent, or study termination; this cohort was closed early due to changes in the first-line standard of care.
  Interventions: Drug: lenvatinib; Drug: Tislelizumab
- Part 2: Urothelial Cancer (UC) Cohort (Experimental): Participants with cisplatin ineligible, systemic therapy naive advanced UC, were to be treated with tislelizumab (400 mg IV Q6W) and lenvatinib (20 mg orally QD). This cohort was closed prior to any participant enrollment based on emerging external data.
  Interventions: Drug: lenvatinib; Drug: Tislelizumab

INTERVENTIONS:
Drug: lenvatinib — Administered at the dose of 20 mg orally, once daily.
Drug: Tislelizumab — 400 mg administered intravenously on Day 1 of each 42-day cycle
  Other Names: BGB-A317

SUMMARY:
This clinical trial evaluated the safety and potential benefits of combining two cancer treatments, tislelizumab and lenvatinib, in Chinese participants with advanced or metastatic cancers, including lung, head and neck, bladder, kidney, and stomach cancer. The study included two parts: the first part assessed how safe the drug combination was, and the second part examined how well it worked.

A small group of participants initially received the drugs to determine the appropriate dose, and if the treatment was well tolerated, additional participants were treated at that dose. Participants remained on the treatment unless their cancer progressed, they experienced serious side effects, or they chose to stop.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants had signed an informed consent form and were able to comply with all study requirements.
2. Participants had a histologically and/or cytologically confirmed diagnosis of advanced solid tumors, which included one of the following types:

   * Non-Small Cell Lung Cancer (NSCLC)
   * Squamous Cell Carcinoma of the Head and Neck (SCCHN)
   * Gastric Cancer (GC)
   * Urothelial Carcinoma (UC)
   * Renal Cell Carcinoma (RCC)
3. Participants had at least one measurable lesion as defined by the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1.
4. Tumor tissue samples (approximately 10 unstained slides) were provided for central laboratory assessment of programmed death-ligand 1 (PD-L1) expression in the NSCLC cohort during the screening period. These samples were also used for retrospective exploratory biomarker analyses related to treatment response and resistance across the NSCLC, SCCHN, UC, or Gastric Cancer (GC) cohorts, in a central or designated test laboratory approved by BeiGene.
5. Participants had an Eastern Cooperative Oncology Group (ECOG) performance of 0 or 1

Key Exclusion Criteria:

1. For participants in the NSCLC cohort, those with active leptomeningeal disease or uncontrolled, untreated brain metastases were excluded. In cohorts other than NSCLC, any participant with known leptomeningeal disease or brain metastases was excluded.
2. Participants who had received prior therapy with lenvatinib, or with antibodies targeting programmed cell death protein 1 (PD-1), programmed death-ligand 1 (PD-L1), programmed death-ligand 2 (PD-L2), or any other agents specifically targeting T-cell costimulatory or immune checkpoint pathways, were excluded.
3. Participants with a history of interstitial lung disease, non-infectious pneumonitis, or any uncontrolled pulmonary conditions (including but not limited to pulmonary fibrosis or acute lung diseases) were excluded.
4. Participants who were unable to swallow capsules, or who had diseases or previous procedures that significantly affected gastrointestinal function such as malabsorption syndrome, surgical resection of the stomach or small bowel, bariatric surgery, symptomatic inflammatory bowel disease, or partial/complete bowel obstruction were excluded.
5. Participants who had experienced clinically significant bleeding (classified as Grade 2 or higher according to the Common Terminology Criteria for Adverse Events [CTCAE]) within 21 days prior to the first dose were excluded.

Note: Additional protocol-defined inclusion and exclusion criteria may have applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-09-18 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2024-07-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Luhe Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - The Peoples Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Cancer Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - Zhejiang Provincial Peoples Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe.
  Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved. BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/

REFERENCES:
- [Background] BGB-A317-212: A Multicenter, Open-label, Phase II Study to Evaluate the Efficacy and Safety of Tislelizumab in Combination With Lenvatinib in Patients With Selected Solid Tumors. Poster No: 2610 presented at ASCO, Chicago, IL, May 31-June 4, 2024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in multiple study centers in China. The first participant dosed was on September 18th, 2021 and the last participant completed on July 10th, 2024. Enrollment began with a run-in phase to assess the safety and tolerability of tislelizumab plus lenvatinib combination therapy. Once the Safety Monitoring Committee confirmed that the combination therapy was tolerable, enrollment into the expansion phase began.
Pre-assignment Details: This study included a safety run-in and expansion phase to evaluate treatment with tislelizumab plus lenvatinib. All participants enrolled in the run-in phase continued into the expansion phase and all participants received the same treatment dose. According to the planned analysis, all enrolled participants were analyzed together (including those who enrolled in the run-in phase) based on tumor type.
Groups:
- Squamous Cell Carcinoma of the Head and Neck (SCCHN): Participants with previously untreated, advanced or metastatic SCCHN received tislelizumab (400 mg administered intravenously [IV] every 6 weeks [Q6W]) in combination with lenvatinib (20 mg taken orally once daily [QD]) until disease progression, start of new anticancer therapy, unacceptable toxicity, withdrawal of consent, or study termination.
- Renal Cell Carcinoma (RCC): Systemic therapy naive participants with advanced or metastatic RCC received tislelizumab (400 mg IV Q6W) plus lenvatinib (20 mg orally QD) until disease progression, start of new anticancer therapy, unacceptable toxicity, withdrawal of consent, or study termination
- Non-Small Cell Lung Cancer (NSCLC): Participants with NSCLC expressing programmed cell death-ligand 1 (PD-L1) in ≥1% of tumor cells (TC ≥1%) and who had not received prior systemic therapy received tislelizumab (400 mg IV Q6W) and lenvatinib (20 mg orally QD) until disease progression, start of new anticancer therapy, unacceptable toxicity, withdrawal of consent, or study termination.
- Gastric Cancer (GC): Participants with advanced GC who had received one prior line of systemic therapy were enrolled to receive tislelizumab and lenvatinib at the RP2D (tislelizumab 400 mg IV Q6W; lenvatinib 20 mg orally QD) until disease progression, start of new anticancer therapy, unacceptable toxicity, withdrawal of consent, or study termination; this cohort was closed early due to changes in the first-line standard of care.
Period: Overall Study
Arm/Group | Squamous Cell Carcinoma of the Head and Neck (SCCHN) | Renal Cell Carcinoma (RCC) | Non-Small Cell Lung Cancer (NSCLC) | Gastric Cancer (GC)
Started | 27 | 23 | 5 | 3
Treated | 27 | 23 | 5 | 3
Enrolled in Safety Run-in Stage | 2 | 0 | 5 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 27 | 23 | 5 | 3
Not completed — Study Completed by Sponsor | 16 | 16 | 3 | 3
Not completed — Death | 11 | 6 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0
Not completed — Miscellaneous. | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set is defined as all participants who received ≥ 1 dose of study drug(s).
Groups:
- Non-Small Cell Lung Cancer (NSCLC): Participants with NSCLC expressing programmed cell death-ligand 1 (PD-L1) in ≥1% of tumor cells (TC ≥1%) and who had not received prior systemic therapy received tislelizumab (400 mg IV Q6W) and lenvatinib (20 mg orally QD) until disease progression, start of new anticancer therapy, unacceptable toxicity, withdrawal of consent, or study termination; this cohort was closed early based on emerging external data.
- Total: Total of all reporting groups
Arm/Group | Squamous Cell Carcinoma of the Head and Neck (SCCHN) | Renal Cell Carcinoma (RCC) | Non-Small Cell Lung Cancer (NSCLC) | Gastric Cancer (GC) | Total
Number analyzed (Participants) | 27 | 23 | 5 | 3 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (10.14) | 62.3 (7.38) | 65.6 (7.92) | 61.3 (9.29) | 62.3 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 1 | 0 | 15
  Male | 19 | 17 | 4 | 3 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 27 | 23 | 5 | 3 | 58
  Other | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety Run-in: Number of Participants With Adverse Events (AEs)
Description: An adverse event refers to any unintended or unfavorable sign, symptom, or condition (including abnormal lab results) that occurs during the study, regardless of whether it is related to the study drug.
  A serious adverse event (SAE) is any untoward medical occurrence that, at any dose:
  * Resulted in death
  * Was life-threatening
  * Required hospitalization or prolongation of existing hospitalization
  * Resulted in disability/incapacity
  * Was a congenital anomaly/birth defect
  * Was considered a significant medical AE by the investigator based on medical judgement.
  A dose-limiting toxicity (DLT) was defined as a Grade 3 or 4 hematologic or nonhematologic toxicity occurring during the DLT assessment window and deemed related to one or more study drugs by the investigator.
Time Frame: From first dose through the end of the safety run-in part, up to 124 days; The DLT observation period was 28 days after first dose.
Population: The Safety run-in set is defined as all participants in the safety run-in stage.
Measure: Count of Participants; unit: Participants
Groups:
- Safety Run-In: Participants with advanced or metastatic unresectable solid tumors were enrolled to receive 400 mg of tislelizumab administered on Day 1 of each 6-week cycle, along with 20 mg of lenvatinib self-administered orally once daily, to determine the recommended Part 2 dose (RP2D).
Arm/Group | Safety Run-In
Number analyzed (Participants) | 7
Participants
  Number of Participants with any TEAEs | 6
  Number of Participants with any SAEs | 4
  Number of Participants with any DLTs | 0

2. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate is defined as the percentage of participants who had a confirmed complete response (CR) or partial response (PR) as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 Tumor assessments.
  CR is defined as the disappearance of all target and non-target lesions and no new lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the first dose up to the primary analysis data cut-off date of 10 October 2023 (maximum time on study was 24.7 months)
Population: Safety Analysis Set: Participants who received ≥ 1 dose of study drug(s) Evaluable Analysis Set: Participants who received ≥ 1 dose of study drug(s), have evaluable disease at baseline, and have ≥ 1 evaluable postbaseline tumor response assessment unless any clinical progressive disease or death occurred before the first postbaseline tumor assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Squamous Cell Carcinoma of the Head and Neck (SCCHN) | Renal Cell Carcinoma (RCC) | Non-Small Cell Lung Cancer (NSCLC) | Gastric Cancer (GC)
Number analyzed (Participants) | 27 | 23 | 5 | 3
Percentage of participants
  Safety Analysis Set | 29.6 [13.8 to 50.2] | 60.9 [38.5 to 80.3] | 20.0 [0.5 to 71.6] | 33.3 [0.8 to 90.6]
  Evaluable Analysis Set: number analyzed (Participants) | 24 | 21 | 5 | 3
  Evaluable Analysis Set | 33.3 [15.6 to 55.3] | 66.7 [43.0 to 85.4] | 20.0 [0.5 to 71.6] | 33.3 [0.8 to 90.6]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from randomization to the first objectively documented disease progression as assessed by the investigator per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1) or death from any cause, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 2
Population: Safety analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Squamous Cell Carcinoma of the Head and Neck (SCCHN) | Renal Cell Carcinoma (RCC) | Non-Small Cell Lung Cancer (NSCLC) | Gastric Cancer (GC)
Number analyzed (Participants) | 27 | 23 | 5 | 3
Months | 6.1 [4.3 to 13.7] | 15.4 [8.4 to NA] — Not estimable due to insufficient number of participants with events | 6.0 [2.5 to NA] — Not estimable due to insufficient number of participants with events | NA [1.4 to NA] — Not estimable due to insufficient number of participants with events

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first documented objective response to documented radiological disease progression as assessed by the investigator using RECIST v1.1, or death from any cause, whichever occurred first. Median DOR was estimated using the Kaplan-Meier method.
  Progressive disease is captured as at least a 20% increase in the sum of diameters of target lesions, using the smallest sum on study as the reference (including the baseline sum if it was the smallest). In addition to the 20% relative increase, the sum also had to show an absolute increase of at least 5 mm.
Time Frame: as for outcome 2
Population: Evaluable Analysis Set. Only participants with best overall response of complete response or partial response confirmed per RECIST v1.1 were included in this analysis,
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Non-Small Cell Lung Cancer (NSCLC): Participants with advanced GC who had received one prior line of systemic therapy were enrolled to receive tislelizumab and lenvatinib at the RP2D (tislelizumab 400 mg IV Q6W; lenvatinib 20 mg orally QD) until disease progression, start of new anticancer therapy, unacceptable toxicity, withdrawal of consent, or study termination; this cohort was closed early due to changes in the first-line standard of care.
- Gastric Cancer (GC): Participants with cisplatin ineligible, systemic therapy naive advanced UC, were recruited to be treated with tislelizumab (400 mg IV Q6W) and lenvatinib (20 mg orally QD). This cohort was closed prior to any participant enrollment based on emerging external data.
Arm/Group | Squamous Cell Carcinoma of the Head and Neck (SCCHN) | Renal Cell Carcinoma (RCC) | Non-Small Cell Lung Cancer (NSCLC) | Gastric Cancer (GC)
Number analyzed (Participants) | 8 | 14 | 1 | 1
Months | 9.6 [2.8 to NA] — Not estimable due to insufficient number of participants with events | NA [10.8 to NA] — Not estimable due to insufficient number of participants with events | 18.5 [NA to NA] — Not estimable for sample size = 1 | NA [NA to NA] — Not estimable due to insufficient number of participants with events and sample size of 1.

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants who demonstrated a confirmed complete response (CR), partial response (PR), or stable disease (SD) as the best overall response, in accordance with the RECIST version 1.1 criteria.
  CR was defined as the disappearance of all target and non-target lesions with no new lesions observed. Any pathological lymph nodes (whether target or non-target) were required to have a reduction in short axis to less than 10 mm.
  PR was defined as at least a 30% decrease in the sum of diameters of target lesions, using the baseline sum of diameters as the reference.
  SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), using the smallest sum of diameters recorded while on study as the reference.
Time Frame: as for outcome 2
Population: Evaluable analysis set and Safety Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Squamous Cell Carcinoma of the Head and Neck (SCCHN) | Renal Cell Carcinoma (RCC) | Non-Small Cell Lung Cancer (NSCLC) | Gastric Cancer (GC)
Number analyzed (Participants) | 27 | 23 | 5 | 3
Percentage of Participants
  Safety Analysis Set | 70.4 [49.8 to 86.2] | 87.0 [66.4 to 97.2] | 100.0 [47.8 to 100.0] | 66.7 [9.4 to 99.2]
  Evaluable Analysis Set: number analyzed (Participants) | 24 | 21 | 5 | 3
  Evaluable Analysis Set | 79.2 [57.8 to 92.9] | 95.2 [76.2 to 99.9] | 100.0 [47.8 to 100.0] | 66.7 [9.4 to 99.2]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to the documented date of death for participants who died on or before the data cutoff date. Median OS was calculated using the Kaplan-Meier method. Data for participants who were alive at the data cutoff date were censored at their last known alive date, defined as either the clinical cutoff date for those still on treatment or the most recent available date confirming they were alive, whichever occurred first.
Time Frame: as for outcome 2
Population: Safety Analysis Set
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Squamous Cell Carcinoma of the Head and Neck (SCCHN) | Renal Cell Carcinoma (RCC) | Non-Small Cell Lung Cancer (NSCLC) | Gastric Cancer (GC)
Number analyzed (Participants) | 27 | 23 | 5 | 3
Month | NA [5.7 to NA] — Not estimable due to insufficient number of participants with events | NA [NA to NA] — Not estimable due to insufficient number of participants with events | NA [NA to NA] — Not estimable due to insufficient number of participants with events | NA [NA to NA] — Not estimable due to insufficient number of participants with events

7. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An adverse event refers to any unintended or unfavorable sign, symptom, or condition (including abnormal lab results) that occurs during the study, regardless of whether it is related to the study drug.
Time Frame: From first dose of study drug to 30 days after last dose, up to the study completion date of 10 July 2024 (up to 32.5 months)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- Squamous Cell Carcinoma of the Head and Neck (SCCHN): Participants with previously untreated, advanced or metastatic SCCHN received tislelizumab (400 mg administered intravenously [IV] every 6 weeks [Q6W]) in combination with lenvatinib (20 mg taken orally once daily [QD]) to evaluate safety and efficacy in the first-line setting.
- Renal Cell Carcinoma (RCC): Systemic therapy naive participants with advanced or metastatic RCC received tislelizumab (400 mg IV Q6W) plus lenvatinib (20 mg orally QD) at the recommended Phase 2 dose (RP2D) to assess clinical benefit in the front-line setting.
- Non-Small Cell Lung Cancer (NSCLC): Participants with NSCLC expressing programmed cell death-ligand 1 (PD-L1) in ≥1% of tumor cells (TC ≥1%) and who had not received prior systemic therapy received tislelizumab (400 mg IV Q6W) and lenvatinib (20 mg orally QD); this cohort was closed early based on emerging external data.
- Gastric Cancer (GC): Participants with advanced GC who had received one prior line of systemic therapy were enrolled to receive tislelizumab and lenvatinib at the RP2D (tislelizumab 400 mg IV Q6W; lenvatinib 20 mg orally QD); this cohort was closed early due to changes in the first-line standard of care.
Arm/Group | Squamous Cell Carcinoma of the Head and Neck (SCCHN) | Renal Cell Carcinoma (RCC) | Non-Small Cell Lung Cancer (NSCLC) | Gastric Cancer (GC)
Number analyzed (Participants) | 27 | 23 | 5 | 3
Participants
  Number of Participants with any TEAEs | 27 | 22 | 5 | 3
  Number of Participants with any SAEs | 17 | 11 | 2 | 2

ADVERSE EVENTS:
Time Frame: All-cause mortality data were collected from randomization through the end of the study (up to 34 months). Serious adverse events (SAEs) and treatment-emergent adverse events (TEAEs) were collected from the date of first study drug administration through 30 days after the last dose (up to 32.5 months).
Arm/Group | Squamous Cell Carcinoma of the Head and Neck (SCCHN) | Renal Cell Carcinoma (RCC) | Non-Small Cell Lung Cancer (NSCLC) | Gastric Cancer (GC)
All-Cause Mortality (participants affected / at risk) | 11/27 | 6/23 | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 17/27 | 11/23 | 2/5 | 2/3
Other Adverse Events (participants affected / at risk) | 27/27 | 21/23 | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Squamous Cell Carcinoma of the Head and Neck (SCCHN) (N=27) | Renal Cell Carcinoma (RCC) (N=23) | Non-Small Cell Lung Cancer (NSCLC) (N=5) | Gastric Cancer (GC) (N=3)
Necrotic lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Squamous Cell Carcinoma of the Head and Neck (SCCHN) (N=27) | Renal Cell Carcinoma (RCC) (N=23) | Non-Small Cell Lung Cancer (NSCLC) (N=5) | Gastric Cancer (GC) (N=3)
Anaemia (Blood and lymphatic system disorders) | 7 (8) | 5 (5) | 1 (1) | 0 (0)
Hypercoagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 4 (6) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cardiac discomfort (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 2 (5) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 10 (16) | 16 (23) | 3 (3) | 1 (1)
Periorbital oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (6) | 2 (2) | 0 (0) | 0 (0)
Alveolar bone defect (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (8) | 5 (5) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Gingival erosion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 7 (11) | 3 (4) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 6 (6) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Facial pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 3 (4) | 1 (1) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 3 (4) | 1 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 5 (6) | 4 (6) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 4 (4) | 10 (12) | 0 (0) | 0 (0)
Fascial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (2) | 2 (2) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Anal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 5 (6) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 2 (2) | 6 (9) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 4 (6) | 0 (0) | 0 (0)
Bile acids increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bilirubin conjugated decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 3 (4) | 7 (18) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Blood corticotrophin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase MB increased (Investigations) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (3) | 5 (6) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (4) | 1 (2) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 2 (3) | 0 (0) | 0 (0)
Granulocyte count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary scan abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 4 (5) | 7 (9) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2) | 3 (5) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (4) | 2 (3) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 8 (9) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 8 (14) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Urine ketone body present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 13 (13) | 13 (15) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (4) | 4 (6) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 6 (7) | 8 (8) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (2) | 6 (7) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (6) | 1 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (14) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 7 (10) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 5 (6) | 1 (1) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5) | 2 (2) | 1 (1) | 0 (0)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyssomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Albuminuria (Renal and urinary disorders) | 2 (4) | 3 (7) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hyperuricosuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IgA nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 7 (12) | 6 (8) | 5 (8) | 1 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scrotal ulcer (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial ulceration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (5) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 (9) | 9 (12) | 3 (5) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 16 (23) | 15 (18) | 4 (5) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT05014828/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT05014828/SAP_001.pdf